CLINICAL TRIAL: NCT06851585
Title: Failure of First-attempt Insertion and Analysis of Practices Related to Peripheral Intravenous Catheters in the Emergency Department: A Prospective Observational Study by the French "Emergency Department Research Initiative" ("Initiatives de Recherche Aux Urgences" IRU) Network
Brief Title: Failure of First-attempt Insertion and Analysis of Practices Related to Peripheral Intravenous Catheters in the Emergency Department:
Acronym: CATHIRU
Status: Completed | Type: Observational
Sponsor: Poitiers University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: CATHIRU
Record Dates: First submitted 2025-02-24; First posted 2025-02-28 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-03

CONDITIONS: Catheterization; Catheterization, Peripheral; Catheters; Vascular Access Devices; Emergency Departments
MeSH Terms: conditions — Emergencies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Cohort of patients with attempted vascular access insertion
  Interventions: Device: CathIRU Cohort

INTERVENTIONS:
Device: CathIRU Cohort — All adult patients requiring a CVP in an emergency department can participate in the study

SUMMARY:
Peripheral intravenous catheters (PIVCs) are essential for the management of hospitalised patients, particularly in emergency departments, where they are used to administer intravenous treatments to more than half of all patients. However, nearly 30% of insertion attempts fail on the first attempt, causing stress and pain for patients and delaying treatment. Despite their importance, PIVC insertion and management practices remain insufficiently standardised and studied, especially in the emergency setting. The CathIRU study aims to address these gaps by investigating the incidence of first-attempt insertion failure and analysing associated practices.

The primary objectives of the study are to estimate the incidence of first-attempt PIVC insertion failure in emergency departments and to identify predictive criteria for difficult vascular access. Secondary objectives include analysing PIVC insertion and management practices, assessing the incidence of unnecessary catheters placed in emergency settings, and evaluating the use of vein access techniques and alternative approaches in cases of failed insertion.

This is a prospective, multicentre observational epidemiological study. It will include 3,000 adult patients requiring a PIVC, recruited over two consecutive days in 70 centres within the IRU network. Data collection will include patient characteristics, insertion site, catheter specifications, insertion techniques, and clinical context.

Inclusion criteria comprise adult patients requiring a PIVC who have provided verbal consent for data collection. Patients with major life-threatening distress or those who had a PIVC inserted in a prehospital setting will be excluded. Data analysis will involve bivariate and multivariate logistic regression to identify risk factors associated with insertion failure and unnecessary catheters, with continuous and categorical data summarised using appropriate descriptive statistics.

The expected benefits of this study include improving PIVC insertion and management practices by enabling early identification of patients at risk of difficult vascular access, reducing complications linked to repeated punctures and delays in diagnostic and therapeutic care, and increasing awareness and training among healthcare professionals in best practices and technologies such as ultrasound guidance. In terms of societal impact, optimising PIVC management is expected to enhance patient care quality, reduce medical costs, and minimise medical waste.

The study is funded by the Société Française de Médecine d'Urgence (SFMU).

ELIGIBILITY:
Inclusion Criteria:

* Adult over 18 years old
* Requiring peripheral vascular access
* Having provided oral consent for data collection

Exclusion Criteria:

* Patient presenting with a state of major life-threatening distress, which may justify the placement of an intraosseous line and/or prevent data collection
* Patient who received vascular access in the prehospital setting
* Patient who has already participated in the study
* Subject not covered by a social security scheme
* Subjects under enhanced protection, namely persons deprived of liberty by a judicial or administrative decision, persons residing in a healthcare or social facility, adults under legal protection (guardianship or curatorship), and patients in emergency situations

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult patients requiring a CVP in an emergency department can participate in the study
Sampling Method: Non-Probability Sample
Enrollment: 4312 (Actual)
Dates: Start 2025-04-03 (Actual); Primary Completion 2025-04-05 (Actual); Study Completion 2025-04-06 (Actual)

PRIMARY OUTCOMES:
Estimate the prevalence of first-attempt PIVC insertion failure | 24 hours
  The prevalence of first-attempt insertion failure will be defined as the number of patients for whom a functional PIVC could not be successfully placed during the first puncture attempt.
  A functional PIVC is defined as one that allows the unrestricted injection of a solution or medication from an infusion line or a flushing syringe. It must be free from complications such as haematoma at the puncture site, extravasation, pain, or arterial reflux.
  We estimate that 20% of patients will experience a first-attempt PIVC insertion failure.

SECONDARY OUTCOMES:
Analyse practices related to the insertion and maintenance of PIVCs | 24 hours
Estimate the percentage of patients presenting with criteria for Difficult Vascular Access | 24 hours
Assess the association between first-attempt insertion failure and the presence of Difficult Vascular Access criteria | 24 hours
Identify the demographic criteria impacting vascular access and predicting failure of insertion at the first attempt | 24 hours
Estimate the prevalence of unnecessary catheters placed in the emergency room | 24 hours
Identify the demographic criteria of centers impacting the incidence of unnecessary catheters placed in emergency departments | 24 hours
Determine the frequency of use of different vein approach techniques | 24 hours
Determine the frequency of use of alternative vascular access in the event of failure of installation | 24 hours

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Poitiers, Poitiers, France, France